CLINICAL TRIAL: NCT04229953
Title: Accuracy of Three /Four-dimensional Ultrasound in Diagnosing Placenta Accreta Spectrum: A Prospective Study
Brief Title: Accuracy of Three /Four-dimensional Ultrasound in Diagnosing Placenta Accreta Spectrum
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hatem AbuHashim (Other)
Responsible Party: Sponsor-Investigator, Hatem AbuHashim, Professor, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: MS.19.05.656
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Placenta Accreta Spectrum
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- US scan with 3D/4D VRU software
  Interventions: Device: US scan with 3D/4D VRU software

INTERVENTIONS:
Device: US scan with 3D/4D VRU software — Every patient will be evaluated by grayscale 2D-ultrasound and color Doppler. Then, a Samsung WS 80A Elite US scanner with 3D/4D VRU software will be used to assess the placental invasion by applying the two modes ("crystal vue" and "realistic vue"). The image analysis will be performed after obtaining the volume dataset. Data will be compared with the intraoperative findings and histopathological confirmation if hysterectomy will be done.

SUMMARY:
The placenta accreta spectrum (PAS) which includes accreta, increta, and percreta represents a significant obstetric challenge. PAS complicates as many as 1 per 500 pregnancies and this risk is increased with prior cesarean deliveries. Antenatal diagnosis of PAS allows for multidisciplinary planning and delivery before the onset of labor and/or vaginal bleeding. This approach has reduced maternal morbidity rates, including less blood loss, fewer transfusion requirements and, intraoperative urologic injuries as well as improve fetal outcome.

Ultrasound evaluation, with grayscale and color Doppler imaging, is the recommended first-line modality for diagnosing PAS. Grayscale ultrasound features suggestive of placenta accreta include an inability to visualize the normal retroplacental clear zone, irregularity and attenuation of the uterine-bladder interface, retroplacental myometrial thickness, presence of intraplacental lacunar spaces, and bridging vessels between the placenta and bladder wall when using color Doppler. Magnetic resonance imaging (MRI) has been used to predict the depth of placental invasion, but it is expensive and often not immediately available.

Recently, a new imaging technique utilizing three-dimensional (3D)/four-dimensional (4D) volume rendering ultrasound (VRU) was proposed as a promising tool for the preoperative diagnosis of placenta previa accerta spectrum. By using "crystal vue" and "realistic vue" volume rendering mode, it could detect 11 out of 12 cases (91.6%) of PAS which was subsequently confirmed during surgery. Accordingly, The aim of this study is to examine the diagnostic performance of 3D/four-dimensional (4D) volume rendering ultrasound (VRU) for placenta previa accerta spectrum in correlation with the clinical (operative) and pathological findings.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in their third trimester
* with a single fetus in the current pregnancy
* a previous delivery by at least 1 cesarean section
* having an anterior placenta previa or anterior low-lying placenta by ultrasound assessment

Exclusion Criteria:

* cases with twin or multiple pregnancies,
* cases with a non-previa placenta or posterior low lying or previa placenta,
* cases without previous deliveries by cesarean section
* cases before the third trimester of pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant females during the third trimester of pregnancy, with a single fetus in the current pregnancy, a previous delivery by at least 1 cesarean section and having an anterior placenta previa or anterior low-lying placenta by ultrasound assessment.
Sampling Method: Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of 3D/4D VRU software | Intra-operative (i.e. during surgery).
  The diagnostic accuracy of 3D/4D VRU software in comparison with the intra operative findings and histopathological confirmation if hysterectomy will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, Study Chair — Faculty of Medicine, Mansoura University; Asmaa Mahran, Principal Investigator — Mahala General Hospital

REFERENCES:
- [Result] Aryananda RA, Akbar A, Wardhana MP, Gumilar KE, Wicaksono B, Ernawati E, Sulistyono A, Aditiawarman A, Joewono HT, Dachlan EG, Parange A, Dekker GA. New three-dimensional/four-dimensional volume rendering imaging software for detecting the abnormally invasive placenta. J Clin Ultrasound. 2019 Jan;47(1):9-13. doi: 10.1002/jcu.22641. Epub 2018 Sep 23. PMID 30246313